CLINICAL TRIAL: NCT03903692
Title: A Comparative Evaluation of a Marine Polysaccharide (MPS) Dressing and a Carboxymethylcellulose (CMC) Dressing on Subjects With Lower Extremity Venous Ulcers
Brief Title: A Comparative Evaluation of a MPS Dressing and a CMC Dressing on Subjects With Lower Extremity Venous Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal stakeholders withdrew funding.
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED-2018-DIV71-026
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-02

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Marine polysaccharide dressing (Experimental)
  Interventions: Device: Marine polysaccharide dressing
- Carboxymethylcellulose dressing (Active Comparator)
  Interventions: Device: Carboxymethylcellulose dressing

INTERVENTIONS:
Device: Marine polysaccharide dressing — The MPS-Ag dressing used in this study has a unique gelling action which helps to remove dead, damaged, and infected tissues from the wound by trapping and removing them later at dressing changes. It is designed to provide intimate contact with the wound for gentle healing. It also contains ionic silver.
  Arms: Marine polysaccharide dressing
Device: Carboxymethylcellulose dressing — The CMC-Ag dressing used in this study incorporates two technologies to help eliminate the key barriers to healing that are exudate, infection, and bioburden. It can be used on chronic and acute wounds that are infected or at risk of infection with varying exudate levels.
  Arms: Carboxymethylcellulose dressing

SUMMARY:
Venous leg ulcers are lower extremity ulcers that develop due to sustained venous hypertension resulting from chronic venous insufficiency. Varicose veins, deep vein thrombosis, poor calf muscle function, arterio-venous fistulae, obesity and history of leg fracture are some of the risk factors for venous ulceration. Numerous dressing types exist to treat these ulcers. This study will compare a marine polysaccharide (MPS) dressing to a carboxymethylcellulose dressing to determine which dressing better manages these wounds with regard to wound size and periwound skin condition. Subjects will be randomized to receive either MPS-Ag dressing or CMC-Ag dressing.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to comply with requirements of this trial protocol
* Voluntarily signed informed consent before any trial related procedures are performed
* Subjects must be able to communicate effectively with study personnel
* Subject has lower extremity venous ulcer wound, as determined by site PI.
* Subject has adequate circulation as determined by biphasic or triphasic Doppler waveform, consistent with adequate blood flow, within three months prior to study enrollment. If monophasic on exam, then non-invasive tests must display Ankle Brachial Index over 0.8 and no worse than mild disease on segmental pressures.
* Subjects should not be allergic to silver (Ag).
* Size of subject's wound is between 1 squared centimeter and 100 squared centimeters.
* Duration of subject's wound is less than 52 weeks.

Exclusion Criteria:

* Subjects who are pregnant, nursing, or planning to become pregnant during the course of the study.
* Subjects who have known allergies to any ingredient(s) in the clinical products used in this study.
* Subjects who do not wish to use products derived from shellfish.
* Subjects with substance use disorder.
* Subjects with active infection or currently receiving antibiotic treatment.
* Subjects who are currently enrolled in another research study which includes investigational treatment and/or medication.
* Subjects judged by the investigator or sub-investigator to be inappropriate as a subject of this study.
* Subject has previous or current systemic disease(s) which, in the judgement of the site PI, is likely to interfere with the study. However, subjects with well-controlled diabetes mellitus (HbA1C < 8.5) shall be permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Valley Vascular Surgery Associates, Fresno, California
  - Central Valley Vein and Wound Center, Selma, California
  - Boston Medical Center, Boston, Massachusetts
  - Covenant Hospital, Saginaw, Michigan
  - Wake Forest Baptist Health, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13 subjects were withdrawn from the study and 6 subjects had unusable data. The analysis was performed on the remaining 43 subjects.
Period: Overall Study
Arm/Group | Marine Polysaccharide Dressing | Carboxymethylcellulose Dressing
Started | 23 | 20
Completed | 23 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Marine Polysaccharide Dressing | Carboxymethylcellulose Dressing | Total
Number analyzed (Participants) | 23 | 20 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.30 (13.14) | 66.75 (11.20) | 65.98 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 12 | 9 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 12 | 15 | 27
  Latino | 10 | 4 | 14
  African American | 0 | 1 | 1
  Asian | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Wound Size From Baseline
Description: Evaluate and compare the percent change in wound size from first to last visit; therefore, percentage change in wound area (mean (t-test) and median (Mann-Whitney U-test)) from first to last visit was calculated for comparison
Time Frame: Baseline to 56 days
Measure: Mean (Standard Deviation); unit: % change in wound area
Arm/Group | Marine Polysaccharide Dressing | Carboxymethylcellulose Dressing
Number analyzed (Participants) | 23 | 20
% change in wound area | 45.61 (36.76) | 56.41 (61.43)

2. Secondary Outcome: Evaluation of Peri-ulcer Skin Assessment Scale
Description: peri-ulcer skin assessment scale is used for assessment. There are 9 systemically items edema, erythema, white atrophy, venous pigmentation, papulovesicular erythema, hyperkeratosis, purpuric patches, telengiectasis, & itching lesions. Each is measured for an extension score 0-4 (0=none; 1=punctual, no extension; 2=local, no extension, does not include total ulcer perimeter; 3=includes total ulcer perimeter, does not include spread beyond; 4=spreads beyond total ulcer perimeter) & severity score from 0-3 (=-none; 1=only detected following examination; 2=clearly apparent; 3=as evident as the wound). The global score is the extension score multiplied by the severity score. Global scores are added together to a total score. Total score scale range 0 - 70 with 0 being the best score and 70 being the worst. All sub-score values, 0 is best score; higher values indicate worsening wounds.
Time Frame: Baseline to 56 days
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Marine Polysaccharide Dressing | Carboxymethylcellulose Dressing
Number analyzed (Participants) | 23 | 20
Score on a scale | 23.5 (18.15) | 24.39 (18.77)

3. Secondary Outcome: Score on a Pain Scale.
Description: Pain was assessed at each dressing change over the course of the study on a scale of 0-10 with 0 being no pain and 10 being the worst pain. The pain score reported was the average of all scores taken at each dressing change for all patients from baseline to 56 days.
Time Frame: Baseline to 56 days
Population: All participants at all dressing changes.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Marine Polysaccharide Dressing | Carboxymethylcellulose Dressing
Number analyzed (Participants) | 23 | 20
Score on a scale | 1.50 (2.46) | 1.65 (2.54)

4. Secondary Outcome: Change in Surface Area of the Dressing
Time Frame: Baseline to 56 days
Population: Percent change was calculated as the area of the dressing at time of application minus the area of the dressing at time of removal, divided by the area of the dressing at time of application, times 100.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Marine Polysaccharide Dressing | Carboxymethylcellulose Dressing
Number analyzed (Participants) | 23 | 20
Percent change | 0.76 (42.11) | 12.65 (48.99)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Marine Polysaccharide Dressing | Carboxymethylcellulose Dressing
All-Cause Mortality (participants affected / at risk) | 0/23 | 1/20
Serious Adverse Events (participants affected / at risk) | 2/23 | 2/20
Other Adverse Events (participants affected / at risk) | 16/23 | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marine Polysaccharide Dressing (N=23) | Carboxymethylcellulose Dressing (N=20)
Serious Adverse Event (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient fell due to pre-existing condition of neuropathy condition not related to her wound. Found not to be related to the products in the study.
Serious Adverse Event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — This SAE was not related to the study products and relevant medical history to this SAE was diabetes, heart burn, deep vein thrombosis (DVT), irregular heartbeat, and hypertension. subject completed final visit.
All-Cause Mortality (Renal and urinary disorders) | 0 (0) | 1 (1) — Death - The unexpected adverse event was end organ failure and not related to study products.
Serious Adverse Event (Gastrointestinal disorders) | 0 (0) | 1 (1) — Subject was admitted to the hospital due to rectal bleeding. Found not to be related to study products.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marine Polysaccharide Dressing (N=23) | Carboxymethylcellulose Dressing (N=20)
Adverse Event (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) — skin conditions found not to be related to study products.
Adverse Event (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Events were found not to be related to study products.
Adverse Event (Surgical and medical procedures) | 8 (8) | 5 (5) — Ablation. not to be related to study products.
Adverse Event (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Found to be related to CoFlex product, not the investigational product.
Adverse Event (Gastrointestinal disorders) | 0 (0) | 3 (3) — Ulcers, found not to be related to study products.
Adverse Event (Infections and infestations) | 1 (1) | 2 (2) — Suspected infections were found not to be related to study products.
Adverse Event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pulmonary congestion with pleural effusion. Found not to be related to study products.
Adverse Event (Renal and urinary disorders) | 0 (0) | 1 (1) — Venaseal and end of organ failure. Found not to be related to study products.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT03903692/Prot_SAP_001.pdf